CLINICAL TRIAL: NCT06614946
Title: Facilitating Effective Coping to Reduce Suicide Risk Following ED Discharge: A Micro-randomized Trial to Develop an Adaptive Text-based Intervention
Brief Title: Improving Coping to Reduce Suicide Risk Following ED Discharge
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ewa Czyz, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00244094; R34MH133057 (NIH)
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Suicidal; Suicide, Attempted; Suicidal Ideation
Keywords: Emergency Department
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation; Emergencies

STUDY DESIGN:
Intervention Model Description: There are 2 arms: ESP only and ESP with text-based program. The ESP with text-based program arm includes twice daily (within-person) randomizations.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic safety plan (ESP) + Text-Based Support (Experimental): Participants who are randomized to this arm will receive ESP during ED care and receive a text-based support program for 4 weeks after discharge, with up to 2 messages per day. The text-based program includes a microrandomized trial (MRT), where participants are randomized twice daily to receive or not receive a message.
  Interventions: Behavioral: Electronic Safety Plan (ESP); Behavioral: Text support
- Enhanced electronic safety plan (ESP) enhanced with 2 reminder text messages with ESP link (Experimental)
  Interventions: Behavioral: Electronic Safety Plan (ESP)

INTERVENTIONS:
Behavioral: Electronic Safety Plan (ESP) — Participants will receive an electronic safety plan in the ED. ESP focuses on developing a personalized coping plan to manage suicidal thoughts and urges.
Behavioral: Text support — Those in the text-based support program will receive up to 2 texts per day for a month with varying levels of tailoring, based on ESP and dynamic personalized feedback.
  Arms: Electronic safety plan (ESP) + Text-Based Support

SUMMARY:
The researchers hope to learn whether an electronic safety plan (ESP) and a supportive text messaging program are feasible and acceptable to adult patients with recent suicidal thoughts or behavior after emergency department (ED) discharge. From this study, the researchers also hope to learn how to best carry out the ESP and text messaging program to improve outcomes for patients after ED discharge.

ELIGIBILITY:
Inclusion Criteria:

Individuals presenting to an ED with either:

1. actual, interrupted, or aborted attempt in the last 4 weeks
2. suicidal ideation within the last week

Exclusion Criteria:

* Severe cognitive impairment or altered mental status (psychosis, manic state)
* Severe aggression/agitation,
* Being admitted or transferred into inpatient care,
* Patient not owning a cell phone with text messaging capability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible individuals who agree to participate | At the time of ED 1 day visit
Completion of the one-month follow-up assessment survey | One month post-discharge from the ED
Completion of the three-month follow-up assessment survey | Three months post-discharge from the ED
Number of withdrawals | Up to 3 months post-discharge from the ED
Percentage of participants who remain active (in text-support condition only) | Up to 28 days post-discharge from the ED
Participant satisfaction with the intervention components | Up to 1 months
  Measured with a modified Client Satisfaction Questionnaire (CSQ).

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Czyz, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No